CLINICAL TRIAL: NCT03956498
Title: Impact of a Sexological Follow-up on the Sexual Function in Patients With Cervix or Vaginal Cancer Treated by Radiotherapy and Brachytherapy
Acronym: FEMINICOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19 GENF 02
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Cervix Cancer; Vaginal Cancer
Keywords: Cervix Cancer; Vaginal Cancer; Sexual function; Brachytherapy; Radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vaginal Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with cervix or vaginal cancer (Other)
  Interventions: Other: Patients with cervix or vaginal cancer treated by radiotherapy and brachytherapy

INTERVENTIONS:
Other: Patients with cervix or vaginal cancer treated by radiotherapy and brachytherapy — * Nurse-led sexological consultations, beginning before brachytherapy and until 2 months after brachytherapy.
  * Questionnaires to be completed by the patient before brachytherapy, 2 months after the end of brachytherapy and 1 year after the end of brachytherapy : Female Sexual Function Index (FSFI), Quality of Life Questionnaire-Core 30 (QLQ-C30), and Quality-of-Life questionnaire cervical cancer module QLQ-CX24.

SUMMARY:
Prospective, monocentric study evaluating the impact of a nurse-led sexological follow-up on sexual function in patients with cervix or vaginal cancer treated by radiotherapy and brachytherapy.

The study procedure will consist of nurse-led sexological consultations, beginning before brachytherapy and until 2 months after brachytherapy.

Evolution of female sexual function and vaginal symptoms will be done through clinical examinations and completion of quality of life and female sexual function questionnaires during radiation oncologist consultation and/or nurse-led sexological consultations until one year after end of brachytherapy.

Study participation of each patient will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Woman diagnosed with cervix or vaginal cancer, for whom a treatment by radiotherapy and brachytherapy has been decided
3. Patient receiving for the first time an utero-vaginal or vaginal brachytherapy at "Institut Universitaire du Cancer de Toulouse - Oncopole"
4. Easter Cooperative Oncology Group (ECOG) Performance Status ≤ 2
5. All patients are eligible, regardless of their relationship status (in couple or not), their sexual orientation, and their hormonal status
6. Patient willing to give informed consent before the study and before performing any study-related procedures
7. Patient affiliated to a Social Health Insurance in France

Exclusion Criteria:

1. Patient not understanding the French language
2. Patient for whom surgical treatment and brachytherapy has been decided
3. Any psychological, familial, sociological or geographical condition that potentially hampers compliance with the study protocol and follow-up after treatment discontinuation schedule
4. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index score (evolution between inclusion and 1 year after brachytherapy) assessed using FSFI (Female Sexual Function Index) Questionnaire | 12 months for each patient

SECONDARY OUTCOMES:
Quality of life assessed using QLQ-C30 questionnaire (Quality of Life Questionnaire-Core 30) | 12 months for each patient
Quality of life specific for cervix cancer assessed using QLQ-CX24 questionnaire (Quality-of-Life questionnaire cervical cancer module) | 12 months for each patient
Vaginal symptoms assessed using NCI-CTCAE version 5 (National Cancer Institute Common Toxicity Criteria for Adverse Events) | 12 months for each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse, France